CLINICAL TRIAL: NCT03130946
Title: Comparison of the Accuracy and Safety of Biopsy in Suspicious Axillary Lymph Nodes With a Crypo-assisted Stick Freeze Biopsy Device or Fine Needle Aspiration
Brief Title: Comparison of Two Types of Biopsy in Suspicious Axillary Lymph Nodes
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruiting rate.
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Houpu Yang, Principal Investigator, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Axbiopsy
Record Dates: First submitted 2017-04-23; First posted 2017-04-27 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Breast Neoplasms
Keywords: breast neoplasms; Ultrasonography, Interventional; Biopsy, Large-Core Needle; Biopsy, Fine-Needle
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Two arm, prospective, open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cryo-assisted core needle biopsy (Experimental): Eligible patients undergo lymph node biopsy with FNA and crpo-assisted stick freeze device sequentially.
  Interventions: Device: Cryo-assisted core needle biopsy; Device: FNA
- Fine needle aspiration alone (Active Comparator): Patients undergo lymph node biopsy with FNA alone.
  Interventions: Device: FNA

INTERVENTIONS:
Device: Cryo-assisted core needle biopsy — Rotational core needle biopsy would be done under local anesthesia. A small incision would be made in the axilla and core needle biopsy be performed using a special cryo-assisted stick freeze device (Cassi II, Scion Medical Technologies, USA). The cytological and histological specimens would be sent for diagnosis.
  Arms: Cryo-assisted core needle biopsy
Device: FNA — FNA would be performed using a 10ml syringe with a 24 gauge needle without anesthesia.

SUMMARY:
Axillary lymph node status is a vital prognostic factor in breast cancer patients and provides crucial information for making treatment decisions. Ultrasound test with subsequent fine needle aspiration (FNA) biopsy in nodes with suspicious features remains the standard of axillary lymph node workup. Insufficient sampling and limited diagnostic accuracy of cytological test compromise the outcome the preoperative lymph node staging strategy especially in patients with intermediate suspicious nodes. This prospective study is to compare the performance of a crpo-assisted core biopsy with FNA.

DETAILED DESCRIPTION:
This prospective study was planned to evaluate the superiority of a core needle biopsy device with a special cryo-assisted rotational design (Cassi II, USA) compared with FNA for biopsy of intermediately suspicious lymph nodes. Eligible patients would be randomized to one of two arms by 1:2 : Core with FNA or FNA alone. The diagnostic accuracy and adverse outcome of core and FNA would be compared.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer.
* With axillary lymph node with thickened cortex.
* Planned for sentinel lymph node biopsy or axillary clearance.

Exclusion Criteria:

* Nodes ultrasonographically normal.
* Nodes with hilar displacement .
* Palpable matted nodes.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of biopsy | Immediate after pathological lymph node stage is available
  True positive rate measures the proportion of positives that are correctly identified by Core needle or FNA

SECONDARY OUTCOMES:
Specificity | Immediate after pathological lymph node stage is available.
  The true negative rate measures the proportion of negatives that are correctly identified.
Sample adequency | Immediate after biopsy specimen is evaluated by pathologists.
  The specimen amount or quality for diagnosis is adequate or not evaluated by pathologists
Adverse effect of surgery | 4 weeks after surgery.
  Hematoma, bleeding need , suture exposure and extrusion.

CONTACTS AND LOCATIONS:
Overall Officials: Shu Wang, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided